CLINICAL TRIAL: NCT05944159
Title: Is the Temporamandibular Joint and Soft Tissue Mobilization Technique Effective in Individuals Diagnosed With Bening Paroxysmal Positional Vertigo?
Brief Title: Temporomandibular Joint and Soft Tissue Mobilisation Techniques on Bening Paroxymal Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Dr, Head of Physiotherapy and Rehabilitation Department, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10354421-2022/06-02
Record Dates: First submitted 2023-04-15; First posted 2023-07-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Soft Tissue Mobilisation; Vestibular Exercises; Physiotherapy; Vertigo, Paroxysmal; Temporomandibular Joint Disorders
Keywords: Bening Paroxymal Positional Vertigo; Temporomandibular Joint Mobilization; Soft Tissue Mobilisation; Vestibular Exrecises; Physiotherapy; Otorhynology
MeSH Terms: conditions — Vertigo; Temporomandibular Joint Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Study Group (n= 20) was recieved Temporomandibular joint ve soft tissue techniques. The techniques were applied 30 minutes once a week for 4 weeks by physiotherapist to the study group.
  Interventions: Behavioral: Study Group
- Control Group (Other): Control group (n=20) was received routin medication therapy was applied. Both groups were asked to do the home exercise program twice a day consisting of vestibular exercise videos sent over whatss app. It was questioned with a phone call once a week whether the exercises were done or not.
  Interventions: Other: Control Group

INTERVENTIONS:
Behavioral: Study Group — Study Group (n= 20) was recieved Temporomandibular joint ve soft tissue techniques. The techniques were applied 30 minutes once a week for 4 weeks by physiotherapist to the study group.
  Arms: Study Group
Other: Control Group — Routin medication therapy was applied to the control group. Both groups were asked to do the home exercise program twice a day consisting of vestibular exercise videos sent over whatss app. It was questioned with a phone call once a week whether the exercises were done or not.
  Arms: Control Group

SUMMARY:
The purpose of this study was to investigated effectiveness of temporamandibular joint and soft tissue mobilization on patients with Benign Paroxysmal Positional Vertigo (BPPV).

DETAILED DESCRIPTION:
Aim: In this study was aimed to investigated effectiveness of temporamandibular joint and soft tissue mobilization on patients with Benign Paroxysmal Positional Vertigo (BPPV). Material and Methods; Dix Hallpike maneuver was administered to all patients to confirm the diagnosis at the initial evaluation. If the Dix Hallpike test was positive, Epley maneuver was applied The patients were randomly divided into 2 groups as study group (n=) and control groups (n= ). Temporomandibular joint ve soft tissue techniques were applied 30 minutes once a week for 4 weeks by physiotherapist. Routin medication therapy was applied to control group. Both groups were asked to do the home exercise program twice a day consisting of vestibular exercise videos sent over whatss app. It was questioned with a phone call once a week whether the exercises were done or not. Patients were evaluated by Dizziness Disability Inventory (DHI) , Dizziness Assessment- Visual Analogue Scale (VAS), Vertigo Symptom Scale-Short Form (VSS) , Beck Anxiety Inventory (BAI) , Vertigo Dizziness Imbalance Questionnaire (VDI) , Tinnitus Disability Scale (TDS), Romberg Posture Test , Tandem Posture Test, Semitandem Tandem Balance Test, Fonseca's Anamnestic Index (FAI) and amount of mouth opening was measured with goniometer before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with positional vertigo,
* Being between the ages of 18-65
* Dix Halpike maneuver test (+),
* Those who volunteered to participate in the study
* Able to read and write.

Exclusion Criteria:

* Findings of acute or chronic infection at the end of ENT examination,
* Considered to have a neurological pathology that causes dizziness,
* Head trauma, history of surgical operation,
* Having lower extremity pain that prevents standing and weight bearing,
* Having a history or symptoms of vestibular system diseases other than BPPV,
* Presence of sudden sensory hearing loss and chronic otitis media,
* Pregnancy,
* The presence of serious cognitive impairment detected by the physician at a level that prevents the tests from being performed,
* Not having the mental level to understand and answer the survey questions,
* Cervical pathologies that may cause dizziness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Dizzness Severity | Baseline - end of the treatment after 4 weeks session
  dizziness severity was determined by Visual Analog Scale (VAS). The patient is asked to evaluate between 0 and 10 points. A score of "0" means no dizziness, a score of "1-4" means mild dizziness, a score of "4-8" means moderate dizziness, and a score of "10" means unbearable dizziness
Vertigo Symptom Scale- Shor Form | Baseline - end of the treatment after 4 weeks session
  It is a 15-item scale that evaluates dizziness, feeling of imbalance, accompanying autonomic disorders and anxiety symptoms in the last 1 month.Each question has values between 0-4 points. The scores of all items will be added together and the total score will be between 0-60 points. High scores indicate serious problems. A total score of 12 points or more indicates a symptom of vertigo. It has 8 items related to vertigo and has a score between 0-32 points, it has 7 items that includes autonomic complaints and has a score of 0-28.
Beck Anxiety Inventory | Baseline - end of the treatment after 4 weeks session
  It were used for to evaluate of anxiety level because of the vertigo. It consists of 21 questions in total.
  0 points: none,
  1. point: mild
  2. points: intermediate,
  3. points: seriously scored. It was classified as mild anxiety symptoms between 8-15 points, moderate anxiety symptoms between 16-25 points, and severe anxiety symptoms between 26-63 points.
Vertigo Dizziness Imbalance Questionnaire (VDI) | Baseline - end of the treatment after 4 weeks session
  The Vertigo-Dizziness-Imbalance Questionnaire is a scale that evaluates the quality of the daily living activities of the problems that patients experience with vertigo and dizzines.Each question has a point value of "4" points if yes, "0" points if no, and sometimes "2" points. In the scoring, 28 points are the limit points for determining physical disability, 36 points for functional and sensory disability.
Tinnitus Disability Scale | Baseline - end of the treatment after 4 weeks session
  The Tinnitus Disability Scale (TDS) was used for the presence and level of balance tinnitus due to vertigo.TDS has 25 questions. The scoring of the answers is "4", "0" and "2" respectively. The lowest score that can be obtained from the scale is 0 and the highest score is 100.
Balance Asssesment | Baseline - end of the treatment after 4 weeks session
  Balance problems due to vertigo were determined by romberg test, tandem and semitandem tests. Romberg Test:In peripheral vestibular pathologies, the direction of the fall is in that direction. For the Tandem and Semitandem tests,It is asked to try to hold the position for 30 seconds with your open eyes closed. The time it can stand is recorded in seconds
The presence of Temporomandibular Joint Disorders | Baseline - end of the treatment after 4 weeks session
  The presence and level of temporomandibular dysfunction was determined by Fonseca's Anamnestic Index (FAI). FAI is a questionnaire consisting of 10 questions and 3 choices. The answers are "yes" (10 points), "sometimes" (5 points), and "no" (0 points). Scoring TMD No signs or symptoms (0-15 points), mild TMD (20-45 points), moderate TMD (50-65 points), and severe TMD (70-100 points)
Mouth opening | Baseline - end of the treatment after 4 weeks session
  amount of mouth opening was measured with goniometer before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayça ARACI, PhD, Study Director — Physiotherapy and Rehabilitation; Dilara GÜLER, Master, Principal Investigator — Physiotherapy and rehabilittaion
Locations (1):
- Alanyaaku, Antalya, Alanya, Turkey (Türkiye)